CLINICAL TRIAL: NCT06951815
Title: The Effect of Hearing Adjustment on the Ease and Effectiveness of Communication, and the Role of Cognitive Resources
Brief Title: The Mental Cost and Burden of Listening
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Sonova AG (Industry)
Responsible Party: Principal Investigator, Stephanie Loukieh, Principle Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-21234-37958
Record Dates: First submitted 2025-04-18; First posted 2025-04-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Quality of Life (QOL); Communication Barriers; Cognitive Performance; Fatigue, Mental
Keywords: Cognitive resource depletion; hearing handicap; hearing loss; listening effort; mental fatigue; ease of communication; sleep efficiency
MeSH Terms: conditions — Mental Fatigue; Hearing Loss

STUDY DESIGN:
Intervention Model Description: The study will include 2 groups of older adult hearing aid candidates, one will receive a hearing aid intervention (the test group) and one will attend an explanation session instead (the control group) and they will be randomly assigned.
  Interested participants will be prescreened over the phone before being invited to the lab for official recruitment. Participants will be invited into the lab if they meet the age requirement (60 or above), get a positive screen in the RHHI-S (6 or above) and meet the condition of having no prior hearing aid experience.
  Participants will be randomly assigned in parallel as enrolment occurs with a biological sex balance. To achieve the randomisation element while still being able to assign as they enrol and maintain biological sex balance, stratified block randomisation will be used with a predetermined random assignment list attached here.
  Both groups will have a pre-test and a post-test.
Masking Description: Concealed allocation prevents the recruiter and data collector from knowing the assignment of each participant before the fitting session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing Aid Group (Experimental): This group will be fitted with hearing aids and will be the intervention group.
  Interventions: Device: Hearing aids programmed to each participant's hearing loss.
- Information Session Control Group (No Intervention): This group will receive an information session during the time that the experimental group receives the hearing-aid fitting about available hearing care solutions.

INTERVENTIONS:
Device: Hearing aids programmed to each participant's hearing loss. — This study is not investigating the efficacy of hearing aids, rather it is investigating the effect of adjusting hearing on cognitive resources, listening effort, and fatigue.
  Arms: Hearing Aid Group

SUMMARY:
This randomised controlled trial aims to test the effect of hearing adjustment using hearing aids, on the ease and effectiveness of communication such as listening effort, fatigue, and sentence recognition in noise, in addition to wellbeing and sleep; and to reveal the role of cognitive resources and sleep efficiency in this relationship.

DETAILED DESCRIPTION:
Participants will be asked to allocate up to 1.5 hours of their time for each of the 3 visits to the lab.

(in fact all activities planned for each visit are estimated to take less than an hour but we are accounting for time to discuss things and allow for questions if needed)

I- Hearing tested:

Once screened over the phone and invited into the lab, all participants will have their hearing tested through PTA thresholds in the lab, done by trained clinical audiologists. This will include standard audiological assessments including otoscopy, obtaining real ear measurements and removing ear wax only if any wax is blocking the ear canal if the participant consents, in order to facilitate the function of the hearing aid so that we avoid wasting the participant's time and study resources.

II- Test Battery:

Both test and control groups will complete a test battery twice: 2 weeks before the hearing aid fitting or the equivalent education session for the control group, and 4 weeks after it. They will also be asked to use a sleep and step tracking device for 2 weeks before, and 4 weeks after the hearing aid fitting / education session. The total number of visits that the participants will be required to make to the lab is 3, during 2 of which they will complete the test battery. The battery is hosted on Gorilla, an experiment platform and presented to them on a university laptop in one of the assigned rooms in the lab.

The test group and the control group will complete the same test battery the same number of times (twice as pre and post-tests).

The test battery is made up of:

1. Demographic questions about age, gender, and whether English is their primary language.
2. The following questionnaires: Pittsburgh Sleep Quality Index - Reduced Morningness-Eveningness Questionnaire - Revised Hearing Handicap Inventory and Screening Tool along with one additional question about whether they have used hearing aids before - WHO-5 questionnaire - Fatigue and Caffeine Screening Questions.
3. Then they will complete the following two groups of tasks which will be counterbalanced:

   * Listening Tasks: Discourse Comprehension Task to Running Speech in Noise (competing speaker) divided into four parts with an Effort visual analogue scale (from NASA-TLX) asking about their effort at each stage - A visual analogue likert scale for Fatigue is requested once before and once after the listening tasks - A speech perception in noise test (multi-speaker babble) where the participants are asked to type whatever they could hear from a sentence spoken in noise (a standardised test that uses AzBio sentences) - A Mental Demand visual analogue scale (from NASA-TLX) is done once at the end of the listening tasks. The listening tasks take around 20 minutes to complete.
   * Cognitive task: Attention Network Test, which takes place for around 20 minutes. It requires the participant to click a keyboard button in relation to the direction of an arrow shown in the centre of the screen over many trials. The arrow is flanked by other arrows that either point in the same direction as the central arrow, or opposite direction, or are straight lines instead of arrows.

All of these assessments in the test battery are either multiple choice questionnaires, or tests where participants press a key on their keyboard in response to visual stimuli on their screen according to a set of instructions. It takes one hour to complete.

III- Intervention:

The test group will be asked to use hearing aids that are fitted specifically for them by clinical audiologists on the research team according to the best practice standards. The hearing aids are state of the art and brand new, provided by SONOVA. The clinical audiologists took part in a training for the specific fitting of SONOVA hearing aids. The control group will not receive this intervention but would take part in an educational session about hearing care solutions instead. The fitting will be customised and every participant will have had ample time to test them before they leave the lab.

SONOVA AG confirms that the hearing aids that this study will trial meet the requirements of the Medical Device Regulation (EU) 2017/745 as well as the Radio Equipment Directive 2014/53/EU, each participant assigned to using the hearing aids can communicate with the research team at any time in case of questions or requests, and will take home all the necessary equipment such as a UK charger and the accessories, and will be trained on how to use them and take care of them. They will also take home a booklet of information for users of the device provided by the manufacturer. The researcher will follow-up with them to make sure that the use of the device is comfortable, see part V below.

IV- Tracking:

Both groups will be asked to use a sleep and step count tracker (in the same device) provided by Activinsights, a device made specifically for clinical trials and research. This device is worn on the wrist like a watch without a screen and it is waterproof, they will be asked to keep it on their wrist day and night for the duration of 6 weeks, 2 of which are before the intervention/education seesion and 4 after. The battery of this device lasts for longer than that so the device will not need any maintenance during that period, it will be given to them fully charged. The data that will be collected from this tracker are step count per day, and sleep efficiency per night, that are calculated based on the device's algorithm for sleep and step tracking.

The actigraph provided by Activinsights called GENEActiv is FDA 510(k) exempt and is a European Class I Medical Device. The participants will take home a leaflet provided by the manufacturer with details about the device, and participants can communicate with the research team at any time if they are experiencing any inconvenience from it. The PI will ensure that the device is working, fully charged, and ready to go before the participant leaves the lab (no charging or maintenance will be required for it).

V- Phone call follow-up:

All participants will be called twice to check in on them regarding their comfort with the device usage, for the test group that entails their use of the hearing aids and the tracker, and for the control group that entails only the tracker. This will include questions about whether they are inconvenienced by the devices, having any negative reactions to anything, and for those using hearing aids additional questions will be based on the Device Oriented Subjective Outcomes DOSO (b) questionnaire which will also be asked at the end of the trial upon returning the hearing aids. This will make sure that the participant receive the support that they need during the period when they are using the devices for the experiment, a script of the call interview questions is attached. The control group participants will be called 3 weeks after the use of the tracker and 5 weeks after, and the test group participants will be called 1 week after hearing aid fitting and 3 weeks after that, and during the hearing aid fitting / education session we will check on all participants' comfort with the sleep tracker in person (forming a third check-up).

VI- Optional EDI Monitoring:

Participants are invited to complete an extra optional online questionnaire to monitor characteristics for the purpose of equality, diversion and inclusion (EDI). As part of the Manchester Biomedical Research Centre (who have advised on the questions asked), we have a commitment to improve access to research participation for diverse communities. In order to do that we need to collect information around characteristics of research participants to identify gaps and develop strategies to deal with these.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 or older
* Hearing aid candidate (hearing loss of an average of 25 dB HL or worse)
* Novice to hearing aids

Exclusion Criteria:

* Younger than 60
* Normal hearing
* Already uses hearing aids

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Subjective Listening-related Mental Fatigue | From enrolment to the end of the trial at 6 weeks
  Subjective listening-related mental fatigue is measured using the Visual Analogue Fatigue Scale at the end of a long listening exercise reworded to reflect listening-related fatigue. It is a one-item scale from 0 to 10, with higher scores indicating more fatigue. This will be measured before the intervention and 4 weeks after, and the analysis will focus on the post-intervention score while controlling for the pre-intervention score.

SECONDARY OUTCOMES:
Subjective Listening-related Effort | From enrolment to the end of the trial at 6 weeks
  Subjective listening-related effort is measured using a one-item, ten-point visual analogue scale from 0 to 10, with higher scores indicating more effort, based on the Effort Subscale of the NASA (National Aeronautics and Space Administration) Task Load Index and reworded to ask about listening-related effort specifically. It is measured as the mean of 4 scales prompted throughout a long listening exercise. This will be measured before the intervention and 4 weeks after, and the analysis will focus on the post-intervention mean score while controlling for the pre-intervention mean score.

OTHER OUTCOMES:
Sentence Recognition in Noise | From enrolment to the end of the trial at 6 weeks
  Performance on sentence recognition in noise is assessed through the number (count) of words that the participant could detect and type into the computer when listening to speech in noise. The correct words would be counted regardless of grammar or spelling mistakes. Higher scores indicate better performance at recognising speech in noise. This will be measured before the intervention and 4 weeks after, and the analysis will focus on the post-intervention score while controlling for the pre-intervention score.
Objective Cognitive Resource Availability | From enrolment to the end of the trial at 6 weeks
  Cognitive resource availability is estimated through measuring the efficiency of the Executive Control Network. The efficiency of the Executive Control Network is measured using RT (Response Time) in milliseconds extracted from the Attention Network Test, which is calculated through the following formula: RT (of all incongruent conditions) - RT (of all the congruent conditions).
  Higher scores indicate less executive control network efficiency and, therefore, less cognitive resource availability. This will be measured before the intervention and 4 weeks after, and the analysis will focus on the post-intervention score while controlling for the pre-intervention score.
Objective Sleep Efficiency | From enrolment to the end of the trial at 6 weeks
  Objective sleep efficiency is measured using a percentage score of time spent asleep divided by time spent in bed averaged over a period of monitoring with an actigraph. The conditions of being asleep and of being in bed are estimated based on actigraphy measurements and algorithms. This will be measured for 2 weeks before the intervention and for 4 weeks after, and the analysis will focus on the post-intervention score while controlling for the pre-intervention score. Scores could range from 0 to 100 with higher scores indicating better sleep efficiency which contributes to better sleep quality.
Subjective Wellbeing | From enrolment to the end of the trial at 6 weeks
  Subjective wellbeing is measured through the "WHO-5" questionnaire provided by the World Health Organisation (WHO). This 5-item questionnaire provides a score from 0 to 100, with higher scores indicating better wellbeing. This will be measured before the intervention and 4 weeks after, and the analysis will focus on the post-intervention score while controlling for the pre-intervention score.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Kluk de-Kort, Doctorate, Study Director — University of Manchester; Antje Heinrich, Doctorate, Study Director — University of Manchester; Josef Schlittenlacher, Doctorate, Study Director — University of Manchester; Stephanie Loukieh, Masters Degree, Principal Investigator — University of Manchester; Raffael Schmitt, Doctorate, Study Director — Sonova AG
Locations (1):
- Manchester Centre for Audiology and Deafness, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Aggregated anonymised data will be shared on an online data registry.